CLINICAL TRIAL: NCT01502917
Title: A Phase I Study of Convection-Enhanced Delivery of 124I-Omburtamab for Patients With Non-Progressive Diffuse Pontine Gliomas Previously Treated With External Beam Radiation Therapy
Brief Title: Convection-Enhanced Delivery of 124I-Omburtamab for Patients With Non-Progressive Diffuse Pontine Gliomas Previously Treated With External Beam Radiation Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Y-mAbs Therapeutics (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11-011
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Brain Cancer; Brain Stem Glioma
Keywords: Brain stem glioma; CNS; MAB 124I-omburtamab; infusion cannula; DIPG; Diffuse Intrinsic Pontine Glioma; 11-011
MeSH Terms: conditions — Brain Neoplasms; Diffuse Intrinsic Pontine Glioma

ARMS (1):
- Radioactive iodine-labeled monoclonal antibody omburtamab (Experimental): This is a therapeutic Phase I study intended to assess the safety of convection-enhanced delivery (CED) of radioimmunotherapy in the treatment of children with diffuse pontine glioma.
  Interventions: Drug: Radioactive iodine-labeled monoclonal antibody omburtamab; Radiation: External Beam Radiotherapy

INTERVENTIONS:
Drug: Radioactive iodine-labeled monoclonal antibody omburtamab — Prior to treatment children will be pre-medicated with super-saturated potassium iodide & liothyronine to prevent thyroid uptake of the therapeutic radioisotopes. The proposed intervention is a surgical procedure using interstitial infusion of the radiolabeled monoclonal antibody 124I-omburtamab into the brain stem tumor. This will be performed by stereotactic placement of a small caliber infusion cannula into the tumor followed by a slow infusion (CED) of 124I-omburtamab. Following treatment, these children will be monitored during inpatient hospitalization with clinical evaluations & PET/CT or PET/MRI scans of the brain & other organs. Clinical observations, intensive care unit monitoring, routine blood & interval imaging studies (MRI & PET/CT or PET/MRI scans) will be performed at predetermined time points. If the PET/CT scan happens to fall on a weekend or holiday, the scan may be done before or after at the discretion of the Study PI. This will not affect dosimetry interpretation.
Radiation: External Beam Radiotherapy — Standard radiation therapy is given 4-6 weeks prior to study entry.

SUMMARY:
The purpose of this study is to test the safety of a new method to treat Diffuse Intrinsic Pontine Glioma (DIPG). The researchers will use "convection-enhanced delivery" (CED) to deliver an agent called 124I-omburtamab. CED is performed during surgery. The study agent is infused through a small tube placed into the tumor in the brain. Many studies have shown this can safely be done in animals but this study is the first time 124I-omburtamab will be given by CED in humans. This will be one of the first times that CED has been performed in the brain stem.

Omburtamab is something called an antibody. Antibodies are made by the body to fight infections and sometimes cancer. The antibody omburtamab is produced by mice and can attack many kinds of tumors. A radioactive substance, 124I-omburtamab, is attached to omburtamab. 124I-omburtamab sticks to parts of tumor cells and can cause the tumor cells to die from radiation. Studies have also been done on humans using 124I-omburtamab to treat other kinds of cancer. Our studies of some DPG and related tumors suggest that omburtamab will bind to the tumor, but the investigators don't know that for sure.

In this study, the researchers want to find out how safe 124I-omburtamab given by CED is at different dose levels. They will look to see what effects (both good and bad) it has on the patient. The dose of 124I-omburtamab will increase for each new group of patients. The procedure has already been safely performed with lower doses and infusion volumes in a number of patients here at MSKCC. The amount they get will depend on when they enter the study. If too many serious side effects are seen with a certain dose, no one will be treated with a higher dose, and some more patients may be treated with a lower dose to make sure that dose is safe.

ELIGIBILITY:
Inclusion Criteria:

* Consensus of diagnosis must be reached by a multidisciplinary pediatric neuro-oncology team by considering both clinical evidence and MRI presentation. Tissue diagnosis is not required.
* The patient must have undergone prior external beam radiotherapy to a dose of 54-60 Gy to the brain stem. At least 4 weeks but no more than 14 weeks must have elapsed from the completion of radiotherapy.
* The patient must be in adequate general condition for study, with Lansky or Karnofsky Performance Score of ≥ 50 at study entry .

Lansky Performance scale will be used for patients ≤16 years of age.

* The patient must be ≥ 2 and ≤ 21 years old.
* Patient must weigh a minimum of 8 kg.

Exclusion Criteria:

* Clinical and/or radiographic (MRI) progression of tumor following external beam radiation therapy.
* Metastatic disease.
* Untreated symptomatic hydrocephalus determined by treating physician.
* AST or ALT > 2x the upper limit of normal.
* Platelets < 100,000/mcL.
* ANC < 1000/mcL.
* Abnormal PT (Inr) >1.5 INR or PTT > 42 sec (may be corrected with FFP, cryoprecipitate, vitamin K, etc).
* Total bilirubin > 2.0 mg/dl.
* Serum creatinine > 1.5x the upper limit of normal for age, or calculated creatinine clearance or nuclear GFR < 70 ml/min/1.73 m2.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 2 years
  Determination that a dose is safe will be made following the treatment of at least 3 but no more than 6 patients at a particular dose level. The dose levels are DL1 (0.25 mCi), DL2 (0.5 mCi), DL3 (0.75 mCi), DL4 (1.0 mCi) DL5 (2.5mCi), DL6 (3.25mCi), DL7 (4.0mCi), DL 7.1(4.0mCi), DL 7.2 (4.0mCi), DL 8 (6.0mCi), DL 9 (8.0mCi), DL 10 (10.0mCi), DL 11 (12.0mCi) ,fallback DL0 (0.125 mCi) FB1 (1.50mCi) and FB2 (2.0mCi). An incidence of dose-limiting toxicity (DLT) in the range of 25% is considered acceptable in this population. A maximum tolerated dose (MTD) will be defined as the dose level below that at which 2 DLTs have occurred.
assess the toxicity profile | 2 years
  Adverse events (toxicity) will be assessed and classified according to the Clinical Terminology Criteria for Adverse Events version 4.0 (CTCAE). Generally, grade 3 toxicities interfere with activities of daily living (ADLs) and grade 4 toxicities are life-threatening. Grade 5 toxicities cause death.

SECONDARY OUTCOMES:
overall survival | 2 years
  Overall survival from the time of diagnosis will be recorded for every patient in this study. Overall survival will be estimated by Kaplan-Meier methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Souweidane, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Souweidane MM, Bander ED, Zanzonico P, Reiner AS, Manino N, Haque S, Carrasquillo JA, Lyashchenko SK, Thakur SB, Lewis JS, Donzelli M, Cheung NV, Larson SM, Kramer K, Pandit-Taskar N, Dunkel IJ. Phase 1 dose-escalation trial using convection-enhanced delivery of radio-immunotheranostic 124I-Omburtamab for diffuse intrinsic pontine glioma. Neuro Oncol. 2025 Sep 17;27(8):2117-2126. doi: 10.1093/neuonc/noaf039. PMID 39969230
- [Derived] Bander ED, Ramos AD, Wembacher-Schroeder E, Ivasyk I, Thomson R, Morgenstern PF, Souweidane MM. Repeat convection-enhanced delivery for diffuse intrinsic pontine glioma. J Neurosurg Pediatr. 2020 Sep 25;26(6):661-666. doi: 10.3171/2020.6.PEDS20280. Print 2020 Dec 1. PMID 32977309
- [Derived] Morgenstern PF, Zhou Z, Wembacher-Schroder E, Cina V, Tsiouris AJ, Souweidane MM. Clinical tolerance of corticospinal tracts in convection-enhanced delivery to the brainstem. J Neurosurg. 2018 Dec 21;131(6):1812-1818. doi: 10.3171/2018.6.JNS18854. Print 2019 Dec 1. PMID 30579270
- [Derived] Souweidane MM, Kramer K, Pandit-Taskar N, Zhou Z, Haque S, Zanzonico P, Carrasquillo JA, Lyashchenko SK, Thakur SB, Donzelli M, Turner RS, Lewis JS, Cheung NV, Larson SM, Dunkel IJ. Convection-enhanced delivery for diffuse intrinsic pontine glioma: a single-centre, dose-escalation, phase 1 trial. Lancet Oncol. 2018 Aug;19(8):1040-1050. doi: 10.1016/S1470-2045(18)30322-X. Epub 2018 Jun 18. PMID 29914796
- [Derived] Ivasyk I, Morgenstern PF, Wembacher-Schroeder E, Souweidane MM. Influence of an intratumoral cyst on drug distribution by convection-enhanced delivery: case report. J Neurosurg Pediatr. 2017 Sep;20(3):256-260. doi: 10.3171/2017.5.PEDS1774. Epub 2017 Jul 7. PMID 28686124
- [Derived] Guisado DI, Singh R, Minkowitz S, Zhou Z, Haque S, Peck KK, Young RJ, Tsiouris AJ, Souweidane MM, Thakur SB. A Novel Methodology for Applying Multivoxel MR Spectroscopy to Evaluate Convection-Enhanced Drug Delivery in Diffuse Intrinsic Pontine Gliomas. AJNR Am J Neuroradiol. 2016 Jul;37(7):1367-73. doi: 10.3174/ajnr.A4713. Epub 2016 Mar 3. PMID 26939629
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/